CLINICAL TRIAL: NCT05618041
Title: The Safety and Efficay Investigation of CAR-T Cell Therapy for Patients With Hematological Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20221019
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoma; Multiple Myeloma
Keywords: CD19,CD20,BCMA; B-ALL/MM/NHL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Autologous T cell injection (Experimental): Patients will be treated with CAR-T cells
  Interventions: Biological: CAR-T Autologous T cell injection

INTERVENTIONS:
Biological: CAR-T Autologous T cell injection — Biological: CAR-T; Drug: Cyclophosphamide,Fludarabine；Procedure: Leukapheresis
  Other Names: CD19 CAR-T; CD20 CAR-T; BCMA CAR-T

SUMMARY:
To evaluate the tolerability and safety of CAR-T technology in patients with relapsed or refractory hematolymphoid malignancies.

DETAILED DESCRIPTION:
Main research purposes:

To evaluate the tolerability and safety of CAR-T technology in patients with relapsed or refractory hematolymphoid malignancies.

Secondary research purposes:

Objective Evaluation of Cytodynamic Characteristics of CAR-T in Different Types of Hematological Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent and be willing and able to comply with the visit, treatment protocol, laboratory examination, and other requirements of the study as specified in the study procedure sheet;
* Diagnosed as recurrent or refractory lymphoma, leukemia or myeloma;
* Tumor cells express targets for CAR-T cell therapy (results: flow cytometry or Immunohistochemical test confirmation);
* Age 14-75 (including threshold), gender unlimited;
* Eastern Cooperative Oncology Group (ECOG) score ≤2;
* HGB ≥ 70g/L (blood transfusion allowed);
* Liver and kidney functions, heart and lung functions meet the following requirements:

  1. Creatinine ≤ 1.5 × ULN;
  2. Left ventricular ejection fraction ≥ 50%;
  3. Blood oxygen saturation>90%;
  4. Total bilirubin ≤ 1.5 × ULN； ALT and AST ≤ 2.5 × ULN;
* For T cell tumor patients, if tumor cells are detected in peripheral blood during screening, flow cytometry should be used to detect that the tumor cell surface immunophenotype is CD4 and CD8 double negative. If the immunophenotype of peripheral blood tumor cells is not double negative for CD4 and CD8, the condition that the proportion of peripheral blood tumor cells is ≤ 1% shall be met;
* Subjects with pregnancy plans must agree to use contraception before entering the study and after the study lasts for six months; If the subject is pregnant or suspected of being pregnant, the investigator shall be informed immediately;
* The subject or guardian understands and signs the informed consent form;
* Expected survival longer than 3 months.

Exclusion Criteria:

* Severe cardiac insufficiency;
* Have a history of severe lung impairment;
* Complicated with other advanced malignant tumors;
* Complicated with severe or persistent infection that cannot be effectively controlled;
* Complicated with severe autoimmune diseases or congenital immune deficiency;
* Active hepatitis (HBV DNA or HCV RNA positive);
* Human immunodeficiency virus (HIV) infection or syphilis infection;
* Have a history of severe allergy to biological products (including antibiotics);
* If there is a history of hematopoietic stem cell transplantation, it should be no more than 6 months before the patient receives allogeneic hematopoietic stem cell transplantation;
* Subjects who received CAR-T therapy or other gene modified cell therapy before screening;
* Conditions that the investigator believes may increase the risk to the subject or interfere with the outcome of the study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-09-06 (Estimated); Study Completion 2027-12-06 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Complete remission (CR) Complete remission with incomplete recovery of blood cells (CRI), positive minimal residual tumor (MRD+) or negative tumor (MRD -) CR/CRI, disease recurrence or progression (PD) were evaluated, and the overall remission rate was ORR=CR+CRI; For drenching Complete remission (CR), partial remission (PR), disease stability (SD) Disease recurrence or progression (PD) was evaluated, and the overall remission rate was ORR=CR+PR; For multiple myeloma Complete remission (CR), partial remission (VGPR, PR), disease stability (SD), disease recurrence or progression (PD) were adopted, Overall remission rate ORR=CR+VGPR+PR;

SECONDARY OUTCOMES:
progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of Senl CAR- T cells in the genomes of PBMC by qPCR method
Cytokine release | 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei w Tian, MD, Study Director — Shanxi Bethune Hospital
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

REFERENCES:
- [Derived] He S, Peng J, Yang X, Meng F, Huang L, Huang L, Tian W, Gao Z, Zhao J, Wang Z, Wei J. Peripheral Blood Smears Distinguish Infective Fever after CAR-T Therapy. Front Biosci (Landmark Ed). 2023 Nov 24;28(11):299. doi: 10.31083/j.fbl2811299. PMID 38062808